CLINICAL TRIAL: NCT02380924
Title: Determination of the in Vivo Recovery and Survival of EryDex (Dexamethasone Sodium Phosphate Encapsulated in Autologous Erythrocytes) in Non-patient Volunteers
Brief Title: Recovery and Survival of EryDex in Non-patient Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Quince Therapeutics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ery51Cr-01-2014
Record Dates: First submitted 2015-02-16; First posted 2015-03-05 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DSP loaded RBC using EryDex System (Active Comparator): Autologous RBC loaded with DSP using the EDS process, and treated RBC are infused to the subject.
  Interventions: Drug: DSP loaded RBC using EryDex System
- Sham treated RBC using the EryDex System (Sham Comparator): Autologous RBC are treated with buffer using the EDS process, and treated RBC are infused to the subject.
  Interventions: Drug: Sham treated RBC using the EryDex System

INTERVENTIONS:
Drug: DSP loaded RBC using EryDex System — Intravenous infusion of 10 mg DSP encapsulated in autologous erythrocytes. Peripheral blood samples are taken over 49 days to determine the 24-hour recovery and survival (T50) of the infused RBC.
  Other Names: EryDex System
  Arms: DSP loaded RBC using EryDex System
Drug: Sham treated RBC using the EryDex System — Intravenous infusion of sham treated autologous erythrocytes. Peripheral blood samples are taken over 49 days to determine the 24-hour recovery and survival (T50) of the infused RBC.
  Other Names: EryDex System
  Arms: Sham treated RBC using the EryDex System

SUMMARY:
This is a randomized, single-blind, single-center, concurrently controlled, exploratory, Phase I study to determine the in vivo kinetics (24-hour post-infusion recovery and T50 survival) of EryDex System (EDS) -processed autologous red blood cells (RBC) in non-patient volunteers. A total of 12 non-patient volunteer subjects will be enrolled and assigned to one of the 2 groups (6 subjects in active arm group, 6 subjects in sham arm group).

DETAILED DESCRIPTION:
EryDex System (EDS) is a combination product used to administer dexamethasone sodium phosphate (DSP) by ex vivo encapsulation in autologous erythrocytes which are re-infused. DSP is dephosphorylated in RBCs to release dexamethasone.

The 12 subjects who meet all of the inclusion/exclusion criteria will be assigned to one of the 2 groups, consisting of 6 subjects each, as follows:

* Group 1 (active drug arm): 15-20 mg DSP loaded in RBC using the EDS.
* Group 2 (sham arm): sham treated autologous RBC using the EDS

One 50±5mL aliquot of blood collected from each subject will be treated using the EDS process (either active drug or sham) and the resultant processed RBCs will be radiolabeled with Chromium-51 (51Cr) for the in vivo kinetic study. A second 10±5mL simultaneously collected sample will be labeled with Technetium-99m (99mTc) to estimate the subject's blood volume. These labeled aliquots will be mixed, and simultaneously infused through a peripheral vein via butterfly or similar catheter (total dose 20-40 μCi). Blood samples will be collected from the subject's contralateral arm immediately pre-infusion and at 5, 7.5, 10, 12.5, 15, 20, and 30 minutes (± 3 min), and on Day 1, 24 hours (±2 h) after completion of infusion. Vital signs will be assessed after the 30-min sample on Day 0 and again on Day 1 before the 24-h sample is collected. Additional blood samples will be collected at 48 (±4 h) and 72 (±4 h) hours and 7 (±1 d) days post-infusion, and then weekly through 49 days post-infusion, with a window of ±2 days for each visit.

ELIGIBILITY:
Inclusion Criteria:

* If female of childbearing potential*, the subject agrees not to donate ova and to use one of 4 methods of contraception from the time of signing the informed consent until 2 months after infusion
* If male, the subject agrees to not donate sperm and to use barrier contraception (e.g., condom with spermicidal cream or jelly) from the time of signing the informed consent until 2 months after infusion
* Physically and mentally healthy, as confirmed by medical history, physical examination, vital signs, clinical laboratory tests, and ECG
* Meets current physical examination guidelines for whole blood donation as set forth by the AABB (Reference Standard 5.4.1A, Standards for Blood Banks and Transfusion Services, 28th edition. Bethesda. TH Carson ed. 2012). Past travel restrictions do not apply for selection of subjects for this study
* Hemoglobin: ≥ 12.5g/dL
* Temperature: ≤ 37.5°C
* Ability to understand the objectives of the trial and comply with the study procedures

Exclusion Criteria:

* Females that are of childbearing potential, pregnant, or are breast-feeding Women of childbearing potential using two forms of birth control (e.g. barrier and hormonal) will be eligible
* Loss/removal of 500 mL or more of blood <4 weeks
* A disability that may prevent the subject from completing all study requirements
* Noncompliance with the study requirements
* Current participation in another clinical study
* Significant occupational exposure to ionizing radiation
* Current or previous neoplastic disease
* History of any impairment of the immunological system
* History of drug or alcohol abuse (<5 years)
* A current diagnosis of severe or unstable cardiovascular disease.
* Any history or current evidence of a cardiac illness as determined by the investigator.
* History or current diagnosis of a psychiatric illness, other than an anxiety disorder, or neurodegenerative disorder.
* History of hemoglobinopathy or G6PD deficiency.
* History of recurrent or chronic infections
* History of tuberculosis
* Have any other significant disease or condition that in the Investigator's opinion would put the subject at risk for participating in the trial, including acute gastric ulcer or diabetes.
* Vital signs persistently outside the following ranges:

  1. Systolic blood pressure <90 or >140 mmHg
  2. Diastolic blood pressure <50 or >90 mmHg
  3. Pulse <50 or >90 bpm. Patients with pulse rates <50 that are otherwise healthy will be eligible for the trial if approved by the Sponsor.
* Any clinically significant ECG abnormality
* Any clinically significant abnormality on standard laboratory examinations, as determined by the Investigator
* Positive serum pregnancy test
* Positive confirmed findings of an infectious disease based on results from the standard blood donor infectious disease screening panel
* Positive results of the drug or alcohol tests at baseline (Day 0 pre-dose) at the unit
* Any previous oral or parenteral steroid use <4 weeks before baseline. Treatment with inhaled or intranasal steroids for asthma or allergies, as well as use of topical steroids will be permitted
* Chronic condition or prior allergic reaction representing a contraindication to the use of dexamethasone or other steroid drugs
* Have participated in any other trial with an investigational drug and received a dose <30 days or 10 half-lives (whichever is greater) from the start of the screening period.
* Requirement for any concomitant medication prohibited by the protocol. Subjects with a history of treatment with oral or depot antipsychotic medication will be excluded
* A drug or treatment known to cause major organ system toxicity during the past year.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
24-hour post transfusion recovery of infused autologous RBCs | 24 hours
  The 24-hour recovery of autologous RBCs loaded with DSP or sham using the EDS will be greater than 75% with 95% confidence. For RBC kinetics and recovery will be reported as mean, 2-sided 95% CI on the mean, standard deviation, minimum and maximum.
Long-term survival of infused autologous RBCs assessed with T50 (Time to disappearance of 50% of the labelled red blood cells from the circulation) | up to 49 days
  For RBC T50 will be reported as mean, 2-sided 95% CI on the mean, standard deviation, minimum and maximum.

SECONDARY OUTCOMES:
Special laboratory tests | up to 49 days
  pH at 37°C, hemolysis, ATP, 2,3-DPG, extracellular potassium, extracellular glucose, extracellular lactate, packed cell volume, RBC morphology and RBC indices. In particular free haemoglobin and and hematuria will be assessed on all defined time points.The measure is a composite outcome

OTHER OUTCOMES:
Safety: Physical exam | up to 49 days
  Physical exam
Safety: Number of abnormal ECGs | up to 49 days
  Number of abnormal ECGs
Safety: Number of adverse events | up to 49 days
  Number of adverse events
Safety: Number of abnormal routine lab values | up to 49 days
  Number of abnormal routine lab values (haematology, chemistry and urinalysis)
Safety: vital signs | up to 49 days
  Vital signs : HR, systolic/diastolic pressure, temperature

CONTACTS AND LOCATIONS:
Overall Officials: Larry J Dumont, PhD, MBA, Principal Investigator — Dartmouth Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States